CLINICAL TRIAL: NCT06910033
Title: CMF SafeTi Fit: Long-term Safety and Performance of CMF Porous Titanium Implants
Brief Title: Long-term Safety and Performance of CMF Porous Titanium Implants
Acronym: CMF SafeTi Fit
Status: Not yet recruiting | Type: Observational
Sponsor: Materialise (Industry)
Responsible Party: Sponsor
Other Study IDs: SMAT011
Record Dates: First submitted 2024-10-31; First posted 2025-04-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Craniofacial Defects
Keywords: Craniofacial Defects; Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Craniomaxillofacial (CMF) porous titanium implant — All patients were treated, between 2016 and 2023, with patient-specific CMF Porous Titanium Implants for facial and/or cranial reconstruction or restoration of bone defects.

SUMMARY:
The goal of this retrospective study is to evaluate the clinical characteristics, efficiency, safety, and long-term performance of craniomaxillofacial (CMF) Porous Titanium Implants within the standard of care across children (0 - <12 years old), adolescent (12 - <22 years old), and adult (≥ 22 years old) populations.

DETAILED DESCRIPTION:
The loss of bone substance or continuity in the cranial and/or facial region can result from trauma, infection, benign or malign tumor resection, and therapeutic side effects (e.g., radiotherapy). CMF Porous Titanium Implants are patient-specific solutions matched with the patient's anatomy to reconstruct bone defects accurately. Following a premarket clinical evaluation and considering long-term risk management, the decision to conduct a retrospective post-market clinical follow-up study was based on identifying possible residual risks and uncertainty about long-term safety and clinical performance that may impact the benefit/risk ratio of the CMF porous titanium devices, thereby ensuring the continued safety and efficacy of these CMF devices.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients of any age are eligible for this study.
* Patients treated with Materialise patient-specific CMF Porous Titanium Implants for facial and/or cranial reconstruction.
* Patients who have followed Standard of Care, as determined in each case by the treating surgeon.

Exclusion Criteria:

* Known hypersensitivity to Titanium at the time of surgery.
* Patients who had or will receive the TMJ Total Arthroplasty System.
* Pregnancy at the time of surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective collection of a minimum of 200 patients that were treated between 2016 and 2023 with patient-specific CMF Porous Titanium Implants for facial and/or cranial reconstruction or restoration of bone defects. All patients included in the study underwent standard visits and follow-up assessments in-hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Last visit success rate of the device after the surgical implantation of Materialise patient-specific CMF Porous Titanium Implants | Last visit (up to 8 years post-implantation)
  Success is defined as follows:
  - The device is securely in place and functional as of the last follow-up or until its removal for reasons unrelated to the device itself.
  Failure is defined as follows:
  * Reoperation without device removal related to the device.
  * Reoperation with device removal related to the device.

SECONDARY OUTCOMES:
Perioperative complications related and unrelated to CMF Porous Titanium Implants | Up to the moment the patient is discharged from the hospital after the procedure (discharge), up to several weeks, depending on defect severity and recovery progress
  Complications related and unrelated to CMF Porous Titanium Implants, including allergic reaction to the anesthetic or titanium (anaphylaxis), complications related to the anesthesia, hematoma, or others.
General post-operative complications up to standard of care (SOC) follow-up | 4 weeks, 3 months, 1 year, 2-3 years, up to 8 years follow-up
  Complications related and unrelated to CMF Porous Titanium Implants, including infection, pain, implant migration, implant exposure, failure of implant, device subsidence, device fracture, diplopia, hematoma, dysesthesia, osteolysis, fistula, wound dehiscence, delayed healing, or others.
Re-intervention rate, implant-related or not | Up to 8 years follow-up
Intraoperative blood loss (mL) | At procedure
  Estimated blood loss by visual inspection or gravimetric method
Technical success of the implantation | At procedure
  Defined by the surgeon, including but not limited to the implantation of the CMF Porous Titanium Implant and guides (if applicable) according to the pre-operative plan without technical difficulties, including design issues, placement issues, planning issues, guides, or others.
Accuracy of the device implantation compared to the pre-operative plan | 4 weeks follow-up
  Accuracy will be quantified by superpositioning the post-operative images with the planning.
Implant migration | 3 months, 1 year follow-up
  Migration will be quantified by calculating the difference between the immediate post-operative and 3-month and 1-year post-operative scans.
Implant time of the device | From surgery up to 8 years
Surgical operation time | At procedure
Total hospital post-operative stay | Up to the moment the patient is discharged from the hospital after the procedure (discharge), up to several weeks, depending on defect severity and recovery progress
  Time of discharge will be registered in eCRF. Post-operative treatment carried out according to the standard practice of the investigational sites will be registered in the eCRF.

CONTACTS AND LOCATIONS:
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No